CLINICAL TRIAL: NCT01914380
Title: PERSEUS - A Prospective Non-interventional Study to Assess the Effectiveness of Aflibercept (Eylea®) in Routine Clinical Practice in Patients With Wet Age-related Macular Degeneration
Brief Title: Investigating the Effectiveness of Eylea in Patients With Wet Age-related Macular Degeneration
Acronym: PERSEUS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 16623; EY1313DE (Other: Company internal)
Record Dates: First submitted 2013-07-23; First posted 2013-08-02 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Wet age-related macular degeneration; Anti-VEGF-Therapy; Observational study
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Patients will be followed-up for 24 months

SUMMARY:
The study aims to investigate the effectiveness of Eylea in patients with wet age-related macular degeneration in routine clinical practice in Germany. The study is purely observational, only data from routine treatment are to be collected. The treatment and treatment conditions are solely at discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with wet wAMD treated with Eylea (in accordance with the local Summary of Product Characteristics, SPC).
* Written informed consent.

Exclusion Criteria:

* Exclusion criteria as listed in the local SPC.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Any concomitant therapy with another agent to treat wet AMD in the study eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with wAMD treated with Eylea. Participants will be recruited from ophthalmological clinics and practices throughout Germany.
  The decision upon treatment is made at the discretion of the attending physician, according to his/her medical practice.
  The medication is prescribed at regular visits to the investigator's office. Commercially available product will be used to treat the patients.
Sampling Method: Non-Probability Sample
Enrollment: 988 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Mean change of visual acuity for the total patient population | Baseline, 12 and 24 months
Mean change of visual acuity for the subgroup of pretreated patients | Baseline, 12 and 24 months
Mean change of visual acuity for the subgroup of non-pretreated patients | Baseline, 12 and 24 months

SECONDARY OUTCOMES:
Monitoring of disease activity | after 12 and 24 months
  Monitoring of disease activity in routine clinical practice setting will be assessed e.g. by determining the o No. of clinical visits (visits for injections) o No. of monitoring visits (visits only for diagnostic purposes, but without injections) o No. of safety visits after the injection (visits only for safety checks after injection) o No. of visits outside the study center o No. of OCT (optical coherence tomography) assessments per patient after 12 and 24 months
Monitoring of treatment patterns | after 12 and 24 months
  same assessment as indicated for "Monitoring of disease activity"
Mean time from indication of Eylea-treatment by the treating physician to start of treatment | after 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany